CLINICAL TRIAL: NCT03601156
Title: Multi-center Study of Preoperative Intraarterial Chemoembolization Combined With Radiotherpy in the Management of Locally Advanced Rectal Cancer
Brief Title: Preoperative Intraarterial Chemoembolization Combined With Radiotherpy in Locally Advanced Rectal Cancer
Acronym: PCAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Dong Wang, chief physician, Third Military Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCAR
Record Dates: First submitted 2015-04-23; First posted 2018-07-26 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2018-07

CONDITIONS: Rectal Cancer
Keywords: rectal cancer; intraarterial chemoembolization; radiotherpy; Oxaliplatin; Tegafur Gimeracil and Oteracil Porassium Capsule
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NATACE-RT (Experimental): Patients receive Oxaliplatin 130mg/m2 intraarterial chemoembolization on day1, and then radiation ( 44 Gy/20 fractions/4 weeks, from day 7 to day 11, day14 to day 18, day 21 to day 25, day 28 to day 32) plus oral S-1 (BSA < 1.25 mm2 receive 80 mg/day; 1.25 mm2 < BSA < 1.5mm2 recive 100 mg/day, BSA>1.5mm2 receive120 mg/day, twice daily, from day 1 to day 28, every 4 weeks)
  Interventions: Device: intraarterial chemoembolization
- NACT-RT (Active Comparator): Patients receive Oxaliplatin 130mg/m2 intravenous chemotherapy on day1, and then radiation ( 44 Gy/20 fractions/4 weeks, from day 7 to day 11, day14 to day 18, day 21 to day 25, day 28 to day 32) plus oral S-1 (BSA < 1.25 mm2 receive 80 mg/day; 1.25 mm2 < BSA < 1.5mm2 recive 100 mg/day, BSA>1.5mm2 receive120 mg/day, twice daily, from day 1 to day 28, every 4 weeks)
  Interventions: Device: intravenous chemotherapy

INTERVENTIONS:
Device: intraarterial chemoembolization
  Arms: NATACE-RT
Device: intravenous chemotherapy
  Arms: NACT-RT

SUMMARY:
Compared to postoperative chemotherapy combined with radiotherapy, preoperative chemotherapy combined with radiotherapy shows higher sphincter preservation rate and lower local recurrence rate in locally advanced rectal cancer. The purpose of this study is to evaluate the response and prognosis of intraarterial chemoembolization and intravenous infusion chemotherapy in patients with rectal T3-T4 and/or N+ rectal cancer before operation.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of rectal cancer, Stage IV.
* Males or females between 18 Years to 75 Years.
* No prior cisplatin-based chemotherapy or radiotherapy.
* Performance status of 0～2 on the ECOG criteria.
* Adequate hematologic (Leukocyte count >= 4,000/uL, neutrophil count >= 1,500/uL, hemoglobin >= 10 g/dL, platelets >= 100,000/uL), hepatic (AST & ALT =< upper normal limit(UNL)x1.5, bilirubin level =< UNLx1.5), and renal (creatinine =< UNL x1.5 or creatinine clearance rate ≥60 ml/min) function.
* Patient can take oral medicine
* Patient compliance that allow adequate follow-up. Informed consent from patient or patient's relative.

Exclusion Criteria:

* Patient with allergic to S-1 or ingredient of Oxaliplatin
* Patient with Peripheral neuropathy
* Diagnosed fibrosis of lung;pulmonary fibrosis or interstitial pneumonia within 28 days.
* Medically uncontrolled serious heart, renal failure, liver failure, hemorrhagic peptic ulcer, paralysis of intestine , ileus, poor controlled diabetes.
* Enrollment in other study.
* Pregnant or breast-feeding.
* Seriously psyche or intelligence problem.
* Inability to comply with protocol or study procedures.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2014-06; Primary Completion 2018-12 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR) | pathologic examination following surgery, at aproximately 9-10 weeks or after preoperative intraarterial chemoembolization plus radiotherpy
  Pathological complete response (pCR) was determined on tumor resection specimens after completion of neoadjuvant therapy, and was defined as no evidence of residual invasive and ductal disease in the rectum and lymph nodes

SECONDARY OUTCOMES:
the Sphincter Preservation Rate | 3 month
Disease-free survival | Following surgery, 5 years
Overall Survival | the first day of treatment to death or last survival confirm date; assesed up to 5 years
Down Staging Rate | Until surgery at 8-9 weeks post chemoradiation plus radiation (which is 4-5 weeks)
Number of Participants with Adverse Events | Until surgery at 8-9 weeks post chemoradiation plus radiation (which is 4-5 weeks)
Number of Postoperative Complication | Until surgery at 8-9 weeks post chemoradiation plus radiation (which is 4-5 weeks)

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Daping Hospital, Third Military Medical University, Chongqing, Chongqing Municipality
  - Chongqing Zhongshan Hospital, Chongqing, Chongqing Municipality
  - Jiangjin Central Hospital, Chongqing, Chongqing Municipality

REFERENCES:
- [Derived] Yang B, Shan J, Feng Y, Dai N, Li M, Chen C, He S, Wang G, Xiao H, Li C, Wang D. Transcatheter rectal arterial chemoembolization with oxaliplatin plus S-1 concurrent chemoradiotherapy can improve the pathological remission rate in locally advanced rectal cancer: a comparative study. Radiat Oncol. 2020 May 6;15(1):94. doi: 10.1186/s13014-020-01540-4. PMID 32375814